CLINICAL TRIAL: NCT01234246
Title: Sexual Dysfunction and the Quality of Sexual Life in Patients With Colorectal Cancer and Their Partners.
Status: Completed | Type: Observational
Sponsor: Tilburg University (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: NL32121.008.10; UVT 2009-4495 (Other Grant/Funding Number: Dutch Cancer Society)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer Patients and Their Partners
Keywords: Colorectal cancer; Sexual function; Sexual dysfunction; Quality of (sexual) life; Partners; Body image; Anxiety (state and trait); Depressive symptoms; Personality
MeSH Terms: conditions — Colorectal Neoplasms; Sexual Dysfunction, Physiological; Coitus; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with colorectal cancer: Patients with colorectal cancer are included
- Partners: Partners of patients with colorectal cancer are included

SUMMARY:
In this project the main focus is on assessing sexual functioning and the quality of sexual life after the treatment of colorectal cancer in patients and their partners.

Patients and their partners complete questionnaires concerning sexual functioning, quality of life, body image, fatigue, anxiety, depressive symptoms, personality factors, and demographic factors. Questionnaires are completed before surgical treatment, 6 weeks, 3 months, 6 months, and 12 months after diagnosis.

The results of this prospective study will give insight in 1) the incidence of sexual problems and the extent patients with colorectal cancer and their partners are bothered by these problems across time, 2) the effect of different treatment modalities on sexual functioning, 3) the relation between sexual problems and quality of life, 4) the determinants of sexual problems and the quality of sexual life adopting the biopsychosocial approach of patients with colorectal cancer who have been treated with surgery, radiation and/or chemotherapy, and more specifically to the role of personality and patient factors and sexual functioning/the quality of sexual life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with colorectal cancer in one of the participating centra, and their partners are asked to participate in this study prior to treatment.
* Patients have to be between 18 and 75 years old.

Exclusion Criteria:

* Disease recurrence at baseline or metastases.
* Poor expression of the Dutch language.
* Dementia.
* History of psychiatric illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer and their partners
Sampling Method: Non-Probability Sample
Enrollment: 1371 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B.L. den Oudsten, PhD, Principal Investigator — Tilburg University; J.A. Roukema, MD, PhD, Principal Investigator — Tilburg University; J. de Vries, PhD, Principal Investigator — Tilburg University
Locations (4):
- Netherlands (4):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Catharina Hospital, Eindhoven
  - St. Elisabeth Hospital, Tilburg
  - TweeSteden Hospital, Tilburg

REFERENCES:
- See also: Website of the Center of Research on Psychology in Somatic Diseases — http://www.uvt.nl/corps
- See also: Website of the Dutch Cancer Society — http://www.kwfkankerbestrijding.nl